CLINICAL TRIAL: NCT03800992
Title: Bad News- Diagnosis: Epilepsy in Childhood
Acronym: Badnews
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02397; ks18Weber
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy in Children
Keywords: SPIKES - a Six-Step Protocol for Delivering Bad News; advisory skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of perception and evaluation of physicians advisory skills per questionnaire — questionnaire according to SPIKES - a Six-Step Protocol for Delivering Bad News to be completed by parents and children (older than eleven)

SUMMARY:
"Bad news" are defined as"any information which adversely and seriously affects an individuals' view of future. Families of chronic ill children are exposed to a high stress load. This project is to investigate the stress burden directly after diagnosis of epilepsy in childhood and coping capabilities in the course of time and how quality of communication at the time of diagnosis effects stress perception and coping behaviour in the following 12 months.

Perceived/ experienced advisory skills of the physician will be assessed by parents and children (older than eleven) on the basis of SPIKES - a Six-Step Protocol for Delivering Bad News.

The subjective perception regarding quality of dialogue in relationship to childrens and their parents quality of life and their coping strategies will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed epilepsy (according to International League Against Epilepsy (ILAE) criteria):
* at least two unprovoked epileptic fits at intervals of at least 24 hours or
* one unprovoked epileptic fit and a recurrence risk of at least 60% or
* epilepsy syndrome

Exclusion Criteria:

* children with intensive care treatment as inpatients
* parents with insufficient German language capabilities
* parents and children with exposure to traumatic events in the past three months that could probably lead to post traumatic distress (loss of a loved person, severe traffic accident, raid, violence, sexual assault, war)

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with newly diagnosed epilepsy at the Universitäts-Kinderspital beider Basel (UKBB), Abteilung Entwicklungs-und Neuropädiatrie, Switzerland and their parents
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
perception of physicians advisory skills with respect to actual distress | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  Evaluation with Six-Step Protocol for Delivering Bad News (SPIKES); enables the physician to fulfill the four most important objectives of the interview disclosing bad news: gathering information from the patient, transmitting the medical information, providing support to the patient, and eliciting the patient's collaboration in developing a strategy or treatment plan for the future.

SECONDARY OUTCOMES:
Change in National Comprehensive Cancer Network (NCCN) thermometer | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  numeric scale ranging from 0 = no distress to 10 = most extreme distress
Change in Stress and Coping Inventory (SCI) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  questionnaire to assess coping strategies; (21 questions asking for stress load assessed by Likert scale; 13 questions asking for stress symptoms assessed by Likert scale)
Change in Adult-Self-Report for Ages 18- 59 (ASR 18-59) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  ASR is a self-report questionnaire for ages 18-59 that assesses behavioral, emotional, and social problems, plus adaptive functioning, personal strengths, and substance use
Change in Stress Coping Style Questionnaire (SVF) 78/78-S | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  questionnaire consists of 78 items divided into 13 scales, each representing a certain way of response to a stressful event: underevaluation, guilt denial, diversion, alternative satisfaction, situation control, reaction control, positive self-instruction, the need for social support, active avoidance, escape tendency, perseveration, resignation, and self-accusation. The levels of the positive and negative strategies are calculated; assessed by Likert scale.
Change in Parenting Stress Index (PSI) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  measure for evaluating the parenting system and identifying issues that may lead to problems in the child's or parent's behavior. Focuses on three major domains of stress: child characteristics, parent characteristics and situational/demographic life stress (48 Items, 12 Subscales)
Change in Pediatric Quality of Life Inventory (Peds-QL) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  standardized, generic assessment instrument that systematically assesses patients' and parents' perceptions of HRQOL in pediatric patients with chronic health conditions,consists of a 15-item core measure of global HRQOL and eight supplemental modules assessing specific symptom or treatment domains
Questionnaire on the assessment of stress and stress management in Childhood and Adolescence Revision (SSKJ 3-8 R) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  assessing composite score: subscale 1 (stress-vulnerability) summed with subscale 3 (stress symptoms and well-being), lower score meaning a better outcome
Child behaviour checklist (CBCL) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  parent-report questionnaire on which the child is rated on various behavioral and emotional Problems in preschool subjects aged 2 to 3 or in subjects between the ages of 4 and 18. It assesses internalizing (i.e., anxious, depressive, and overcontrolled) and externalizing (i.e., aggressive, hyperactive, noncompliant, and undercontrolled) behaviors. Several subareas were measured including social withdrawal, somatic complaints, anxiety and depression, destructive behavior, social problems, thought problems, attention problems, aggressive behavior, and delinquent behaviors.
Pediatric Quality of Life Inventory (PedsQL 4.0) | 1 -2 days and 6 months and 12 months after first communication of epilepsy diagnosis to parents and child
  The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL Disease-Specific Modules. The PedsQL 4.0 Generic Core Scales consist of 23 items applicable for healthy school and community populations, as well as pediatric populations with acute and chronic health conditions; The PedsQL 4.0 Generic Core Scales instrument consists of the following 4 domains: (1) physical functioning, (2) emotional functioning, (3) social functioning, and (4) school functioning. It includes formats for typically developing children and adolescents 2 to 18 years old (parent-proxy report) and 5 to 18 years old (self-report); Higher scores indicate better HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weber, Prof. Dr., Principal Investigator — Universitäts-Kinderspital beider Basel UKBB
Locations (1):
- Universitäts-Kinderspital beider Basel UKBB, Basel, Switzerland